CLINICAL TRIAL: NCT00817440
Title: Effects of Fasting and Exercise on Insulin and GH Signaltransduction in Muscle and Fat
Acronym: FEIGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Mikkel Vendelbo MD, endokrinologiskforskningslaboratorium M, Aarhus sygehus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16.12.2008
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: growth hormone insulin signaltransduction signalpathways; growth hormone and insulin signalpathways
MeSH Terms: interventions — Exercise; Angptl4 protein, mouse

ARMS (3):
- Control (No Intervention): control: muscle and fat biopsies and basal aminoacid and glucose turnover
- Exercise (Experimental): 1 hour ergometer cycling on 65% of Vo2max, and then the same as arm 1.
  Interventions: Other: Exercise
- Fasting (Experimental): 3 days of fasting and then the same as arm 1
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Exercise — 1 hour ergometer cycling on 65% of Vo2max, and then the same as arm 1.
  Arms: Exercise
Other: Fasting — 3 days of fasting and then the same as arm 1
  Arms: Fasting

SUMMARY:
Hypothesis: under fasting there will primarily be an activation of growth hormone(GH) signalpathways and a inhibition of insulin signalpathways, and the opposite will happen under physical activity.

Primarily we will investigate markers for GH and insulin signaltransduction in muscle- and fat-biopsies after fasting for 72 hours and after 1 hour of ergometer-cycling at 65% Vo2max.

In addition to this we will investigate the effect of fasting and exercise on the velocity of carbamide synthesis, aminoacid rate of turnover and glucose rate of turnover.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* Body mass index (BMI) 20-26
* age 18-45 years

Exclusion Criteria:

* any kind of disease
* any use of medicine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Growth hormone and insulin signal pathways | 30 min

SECONDARY OUTCOMES:
aminoacid and glucose turnover | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus sygehus, Aarhus, Jylland, Denmark